CLINICAL TRIAL: NCT02058121
Title: Randomised Controlled Trial With Acceptance and Commitment Therapy (ACT) for Patients With Eating Disorders - a Manualised Group Therapy to Enhance Body Acceptance
Brief Title: An ACT Group Intervention for ED-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Sanna Aila Gustafsson, Med.dr, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/294
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Eating Disorder
Keywords: Eating disorders; Acceptance and Commitment Therapy; Body image
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — ACT is provided in 12 weekly two hour long sessions in a group setting
  Arms: Acceptance and Commitment Therapy
Behavioral: Treatment as usual — Treatment as usual contains different interventions available at the clinic, such as individual therapy, group therapy, or contact with a physician, dietician and/or physiotherapist.
  Arms: Treatment as usual

SUMMARY:
The purpose of this study was to test if an ACT group intervention focusing on body image reduces eating disorders symptoms and reduces care consumption in patients treated at a specialised eating disorder unit.

DETAILED DESCRIPTION:
The study is an RCT in which the ACT-intervention is compared to treatment as usual. The trial started in 2010, and randomisation of patients continued until 2014, and follow-ups was completed in 2016.

According to analysis of power, a total of 120 patients needed to be included, 60 in each arm. Patients eligible for the interventions were invited to participate after their clinician reported them to the head investigator. The head investigator sent a letter to the patients with information on the study. The clinician then asked the patient if the letter had been read. If the patient wanted to participate, he/she was invited to an information and assessment meeting. The head investigator made sure that the patient understood the information, and what each study arm might mean for the patient when participating. Consent to participate was collected both verbally and in writing. At this meeting the patient received an envelope which contained the randomisation outcome. The patient then received information regarding the continued treatment according to which research arm he/she was to participate in.

The participants randomised to treatment as usual continued with the treatment as planned before enrolment.

Participants in the intervention arm started the group intervention consisting of 12 sessions over a period of three to four months. The intervention also included one individual meeting with the group-leaders before and one after the intervention. The intervention is a manualised application of the book "Lev med din kropp" [Live with your body]. Participants who were in need of further care after the intervention were offered continued treatment accordingly at the clinic.

If a participant chose to terminate the intervention, or deteriorated during the intervention to the point that other treatment was needed, further treatment was agreed upon in dialogue with the patient. If needed, further assessment and physical examination was conducted in accordance to the clinics standard procedures.

Data was collected at four times for all participants. At treatment start and end, and follow-up at 12 and 24 months after inclusion. At each time, the participants were prompted to fill in five different self-assessment forms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an eating disorder according to DSM-IV (APA, 1994)
* Enrolled as a patient at Eriksbergsgarden, a clinic in Sweden offering specialized care for patients with an eating disorder
* Attained a somewhat regular eating pattern consisting of at least three meals per day

Exclusion Criteria:

* Having physical or psychiatric complicating factors of such severity that these conditions needed to be addressed during the treatment period (12 weeks).

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptoms | 24 months follow up
  Assessed through the Eating Disorder Examination-Questionnaire (EDE-Q). The EDE-Q consists of 28 questions assessing eating disordered symptoms for the past 28 Days. A global score is calculated based on 22 of the items, ranging from 0-6. The 22 items can be divided into four subscales, assessing eating restraint, eating concern, shape concern and weight concern, also in the range of 0-6. A higher score indicates more severe eating disordered symptoms.

SECONDARY OUTCOMES:
Changes in Mindful awareness | 24 month follow up
  Assessed through the Mindful Attention Awareness Scale (MAAS). The MAAS consists of 15 questions, ranging from 1 to 6. A global score is calculated where higher scoring indicates more mindful awareness.
Measure of body shape preoccupations. | 24 months
  Assessed through the Body Shape Questionnaire (BSQ), a short Swedish version consisting of 8 questions. A total score is calculated, ranging from 8 to 48, where higher scoring indicates more severe concerns.
Measurement of body checking | 24 months
  Assessed through the Body Checking Questionnaire (BCQ). The BCQ consist of 23 questions ranging from 1 to 5. A global score is calculated ranging from 23 to 115, where a higher scoring indicates more frequent use of behaviours related to a negative body image.
Measure changes in self-concept | 24 months
  Assessed through the Self-Concept Questionnaire (SCQ). The SCQ consists of 30 questions ranging from 0 to 7. A global score is calculated where higher scorings indicates a higher self-esteem.

OTHER OUTCOMES:
Differences in amount of healthcare received after treatment intervention | 24 months
  Assess the amount of received healthcare at the eating disorder clinic in terms of amounts of sessions after the intervention endpoint, and at end of follow-up.
The participants opinions regarding the intervention | 24 months
  After last follow up participants are asked to participate in a qualitative interview, with focus on what was helpful and not in the intervention, according to the participants own reflections

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Gustafsson, PhD, Principal Investigator — Psychiatric research centre, Orebro County Counsil
Locations (1):
- Eriksbergsgarden, Orebro County Counsil, Örebro, Orebro County Counsil, Sweden

REFERENCES:
- [Derived] Fogelkvist M, Parling T, Kjellin L, Gustafsson SA. A qualitative analysis of participants' reflections on body image during participation in a randomized controlled trial of acceptance and commitment therapy. J Eat Disord. 2016 Dec 12;4:29. doi: 10.1186/s40337-016-0120-4. eCollection 2016. PMID 27999670